CLINICAL TRIAL: NCT03751124
Title: An International Phase 3 Double-Blind, Placebo-Controlled, Randomized Withdrawal Study of Relugolix With Estradiol and Norethindrone Acetate in Women With Heavy Menstrual Bleeding Associated With Uterine Fibroids
Brief Title: Study of Relugolix With Estradiol and Norethindrone Acetate in Women With Heavy Menstrual Bleeding Associated With Uterine Fibroids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Myovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MVT-601-035; 2018-001368-43 (EudraCT Number)
Record Dates: First submitted 2018-11-13; First posted 2018-11-23 (Actual); Results first posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-05

CONDITIONS: Uterine Leiomyoma; Uterine Fibroids
Keywords: Heavy menstrual bleeding; Menorrhagia; Uterine Fibroids; Uterine Leiomyoma
MeSH Terms: conditions — Myofibroma; Leiomyoma; Menorrhagia | interventions — relugolix; estradiol, norethindrone drug combination

STUDY DESIGN:
Intervention Model Description: Randomized withdrawal following an open-label extension to a randomized controlled parent study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Relugolix plus E2/NETA (Experimental): Relugolix 40 mg co-administered with estradiol (1.0 mg) and norethindrone acetate (0.5 mg) for up to 52 weeks.
  Interventions: Drug: Relugolix; Drug: Estradiol/norethindrone acetate
- Placebo tablets and capsules (Placebo Comparator): * Placebo for relugolix co-administered with placebo for E2/NETA for up to 52 weeks or until heavy menstrual bleeding returns.
  * Retreatment with open-label relugolix with E2/NETA will be offered if heavy menstrual bleeding returns.
  Interventions: Drug: Placebo for relugolix; Drug: Placebo for E2/NETA

INTERVENTIONS:
Drug: Relugolix — Relugolix 40 mg tablet administered orally once daily
  Other Names: TAK-385
  Arms: Relugolix plus E2/NETA
Drug: Estradiol/norethindrone acetate — Capsule containing co-formulated tablet of estradiol 1.0 mg and norethindrone acetate 0.5 mg administered orally once daily
  Other Names: E2/NETA; Low-dose hormonal add-back
  Arms: Relugolix plus E2/NETA
Drug: Placebo for relugolix — Placebo tablet administered orally once daily and manufactured to match the relugolix tablet in size, shape, color, and odor
  Arms: Placebo tablets and capsules
Drug: Placebo for E2/NETA — Placebo capsule administered orally once daily and designed to match the E2/NETA capsule in size, shape, color, and odor
  Arms: Placebo tablets and capsules

SUMMARY:
The objectives of this randomized withdrawal study are to evaluate the long-term efficacy and safety of the combination of relugolix, estradiol (E2) and norethindrone acetate (NETA), once daily, for up to 104 weeks in patients with uterine fibroids who have completed a total of 52 weeks of treatment, including a 24-week treatment period in a parent study (study MVT-601-3001 or MVT-601-3002) and a 28-week treatment period in the open-label extension study (MVT-601-3003), and who meet the definition of responder, defined as a patient who demonstrates a menstrual blood loss of < 80 mL and at least a 50% reduction from parent study baseline menstrual blood loss volume on the alkaline hematin analysis of the feminine products returned at Week 48 in the extension study.

DETAILED DESCRIPTION:
This randomized withdrawal study is an international phase 3 double-blind, placebo-controlled study that will enroll eligible patients with uterine fibroids who have completed the 24-week treatment period in a parent study (MVT-601-3001 or MVT-601-3002) and the 28-week treatment period of the open-label extension study (MVT-601-3003). When including treatment during the parent study and the extension study, patients completing this randomized withdrawal study will have received up to a total of 104 weeks of treatment with relugolix.

Approximately 360 women with heavy menstrual bleeding associated with uterine fibroids completing the extension study with a response to treatment will be eligible to participate in this study. A responder is defined as a patient who demonstrates a menstrual blood loss of < 80 mL and at least a 50% reduction from parent study baseline menstrual blood loss volume on the alkaline hematin analysis of the feminine products returned at Week 48 in the extension study.

Screening procedures will be done on the same day as the Week 52 visit for the extension study. This visit will be referred to as the "Week 52/Baseline visit." When the Week 52/Baseline procedures in the extension study have been completed, the investigator will assess patient eligibility for participation in this study. The eligibility assessment will be based on data available at the Week 52/Baseline visit.

Patients will be asked to provide feminine products for alkaline hematin analysis at each visit until the analysis confirms the return of heavy menstrual bleeding. The patients will then be offered retreatment with open-label relugolix with E2/NETA with the onset of the next menses. They will resume collection of feminine products for alkaline hematin analysis until two consecutive analyses confirm resolution of heavy menstrual bleeding (menstrual blood loss of < 80 mL). Safety will be assessed throughout the study by monitoring adverse events, vital signs, physical examinations, clinical laboratory tests, and assessments of bone mineral density.

ELIGIBILITY:
Inclusion Criteria:

1. Completed the open-label extension study (MVT-601-3003).
2. Is a responder: Has a menstrual blood loss of < 80 mL AND at least a 50% reduction from the parent study Baseline based on the results of the alkaline hematin testing performed on the feminine products returned at the Week 48 visit of the extension study.
3. Is not expected to undergo gynecological surgery or ablation procedures for uterine fibroids within the study period

Exclusion Criteria:

1. Has undergone myomectomy, ultrasound-guided laparoscopic radiofrequency ablation, or any other surgical procedure for fibroids, uterine artery embolization, magnetic resonance guided focused ultrasound for fibroids, or endometrial ablation for abnormal uterine bleeding at any time during the Parent study or extension study.
2. Has a weight that exceeds the weight limit of the dual-energy x-ray absorptiometry (DXA) scanner
3. Has developed any contraindication to treatment with estradiol or norethindrone acetate
4. Is currently pregnant or lactating, or intends to become pregnant during the study period
5. Met a withdrawal criterion in the open-label extension (OLE) study.

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 229 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-10-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (95):
- United States (65):
  - Birmingham, Birmingham, Alabama
  - Mesa, Mesa, Arizona
  - Tucson, Tucson, Arizona
  - Canoga Park, Canoga Park, California
  - Huntington Beach, Huntington Beach, California
  - La Mesa, La Mesa, California
  - Los Angeles, Los Angeles, California
  - Norwalk, Norwalk, California
  - San Diego, San Diego, California
  - Denver, Denver, Colorado
  - Lakewood, Lakewood, Colorado
  - Aventura, Aventura, Florida
  - Clearwater, Clearwater, Florida
  - Deland, DeLand, Florida
  - Ft. Lauderdale, Fort Lauderdale, Florida
  - Fort Myers, Fort Myers, Florida
  - Jacksonville, Jacksonville, Florida
  - Jupiter, Jupiter, Florida
  - Margate, Margate, Florida
  - Miami, Miami, Florida
  - Orlando, Orlando, Florida
  - Oviedo, Oviedo, Florida
  - Sarasota, Sarasota, Florida
  - Tampa, Tampa, Florida
  - United States, Florida, West Palm Beach, Florida
  - West Palm Beach, West Palm Beach, Florida
  - Weston, Weston, Florida
  - Atlanta, Atlanta, Georgia
  - Augusta, Augusta, Georgia
  - College Park, College Park, Georgia
  - Dacatur, Decatur, Georgia
  - Duluth, Duluth, Georgia
  - Norcross, Norcross, Georgia
  - Savannah, Savannah, Georgia
  - Smyrna, Smyrna, Georgia
  - Chicago, Chicago, Illinois
  - Oak brook, Oak Brook, Illinois
  - Shawnee, Shawnee Mission, Kansas
  - Covington, Covington, Louisiana
  - Marrero, Marrero, Louisiana
  - Metairie, Metairie, Louisiana
  - Baltimore, Baltimore, Maryland
  - Towson, Towson, Maryland
  - Canton, Canton, Michigan
  - Detroit, Detroit, Michigan
  - Las Vegas, Las Vegas, Nevada
  - Lawrenceville, Lawrenceville, New Jersey
  - Williamsville, Williamsville, New York
  - Durham, Durham, North Carolina
  - Raleigh, Raleigh, North Carolina
  - Winston Salem, Winston-Salem, North Carolina
  - Cincinnati, Cincinnati, Ohio
  - Bluffton, Bluffton, South Carolina
  - Charleston, Charleston, South Carolina
  - Columbia, Columbia, South Carolina
  - Chattanooga, Chattanooga, Tennessee
  - Memphis, Memphis, Tennessee
  - Dallas, Dallas, Texas
  - Houston, Houston, Texas
  - Longview, Longview, Texas
  - San Antonio, San Antonio, Texas
  - Webster, Webster, Texas
  - Norfolk, Norfolk, Virginia
  - Richmond, Richmond, Virginia
  - Spokane, Spokane, Washington
- Brazil (5):
  - Porto Alegre, Porto Alegre, Rio Grande do Sul
  - São Bernardo do Campo, São Bernardo do Campo, São Paulo
  - Sao Paulo, São Paulo, São Paulo
  - Porto Alegre, Porto Alegre
  - São Paulo, São Paulo
- Chile (3):
  - Providencia, Providencia
  - San Ramon, San Ramón
  - Santiago, Santiago
- Czechia (3):
  - České Budějovice, České Budějovice
  - Olomouc, Olomouc
  - Pisek, Písek
- Hungary (5):
  - Kecskemét, Kecskemét, Bács-Kiskun county
  - Debrecen, Debrecen
  - Gyula, Gyula
  - Nyíregyháza, Nyíregyháza
  - Szentes, Szentes
- Italy (4):
  - Catanzaro, Catanzaro
  - Roma, Roma
  - SIENA, Siena
  - Torino, Torino
- Poland (5):
  - Szczecin, Szczecin, West Pomeranian Voivodeship
  - Bialystok, Bialystok
  - Katowice, Katowice
  - Poznan, Poznan
  - Warszawa, Warsaw
- South Africa (5):
  - Bloemfontein, Bloemfontein, Free State
  - Centurion, Centurion, Gauteng
  - Cape Town, Cape Town, Western Cape
  - Durban, Durban
  - Roodepoort, Roodepoort

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Hendy A, Venturella R, Arjona Ferreira JC, Li Y, Soulban G, Wagman RB, Lukes AS. LIBERTY randomized withdrawal study: relugolix combination therapy for heavy menstrual bleeding associated with uterine fibroids. Am J Obstet Gynecol. 2023 Dec;229(6):662.e1-662.e25. doi: 10.1016/j.ajog.2023.08.030. Epub 2023 Sep 2. PMID 37666383

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed the long-term extension study with a response to treatment, signed the informed consent form, and met all eligibility criteria were enrolled in the study.
Pre-assignment Details: One participant in the placebo group was randomized in error and did not receive treatment, therefore, not included in the modified intent-to-treat (mITT) population.
Groups:
- Relugolix Plus Estradiol (E2) /Norethindrone Acetate (NETA) (Group A): Relugolix 40 mg co-administered with E2 (1 mg) and NETA (0.5 mg) for up to 52 weeks.
- Placebo (Group B): Relugolix placebo co-administered with E2 and NETA placebo for up to 52 weeks.
Period: Overall Study
Arm/Group | Relugolix Plus Estradiol (E2) /Norethindrone Acetate (NETA) (Group A) | Placebo (Group B)
Started | 115 | 114
Received at Least 1 Dose of Study Drug | 115 | 113
Completed | 89 | 86
Not Completed | 26 | 28
Not completed — Adverse Event | 4 | 3
Not completed — Protocol Deviation | 0 | 1
Not completed — Lost to Follow-up | 6 | 4
Not completed — Withdrawal by Subject | 6 | 8
Not completed — Lack of Efficacy | 1 | 1
Not completed — Pregnancy | 0 | 1
Not completed — Other | 9 | 9
Not completed — Participants who did not receive any study drug | 0 | 1

BASELINE CHARACTERISTICS:
Population: mITT population: all participants randomized to treatment who had taken at least one dose of study treatment (relugolix plus E2/NETA or placebo).
Groups:
- Relugolix Plus E2/NETA (Group A): Relugolix 40 mg co-administered with E2 (1 mg) and NETA (0.5 mg) for up to 52 weeks.
- Total: Total of all reporting groups
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B) | Total
Number analyzed (Participants) | 115 | 113 | 228
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (5.58) | 44.2 (4.39) | 43.8 (5.04)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 115 | 113 | 228
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 29 | 58
  Not Hispanic or Latino | 85 | 84 | 169
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Number of participants based on their race.
  Participants
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 1 | 1 | 2
    Black or African American | 49 | 57 | 106
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    White | 63 | 52 | 115
    Other | 1 | 2 | 3
    Multiple | 0 | 0 | 0
    Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Hungary | 4 | 8 | 12
  United States | 74 | 74 | 148
  Czechia | 2 | 1 | 3
  Brazil | 5 | 2 | 7
  Poland | 14 | 12 | 26
  Italy | 6 | 3 | 9
  South Africa | 7 | 6 | 13
  Chile | 3 | 8 | 11
Bone Mineral Density (BMD) at Week 52/Baseline [Mean (Standard Deviation); unit: g/cm^2] — Population: The data was reported for participants analyzed for each parameter.
  g/cm^2
    Lumbar Spine (L1-L4): number analyzed (Participants) | 111 | 112 | 223
    Lumbar Spine (L1-L4) | 1.18 (0.173) | 1.20 (0.147) | 1.19 (0.160)
    Total hip: number analyzed (Participants) | 111 | 110 | 221
    Total hip | 1.04 (0.151) | 1.04 (0.140) | 1.04 (0.145)
    Femoral neck: number analyzed (Participants) | 111 | 110 | 221
    Femoral neck | 0.97 (0.186) | 0.97 (0.164) | 0.97 (0.175)
Mean Menstrual Blood Loss (MBL) Volume at Week 52/ Baseline [Mean (Standard Deviation); unit: mL] | 8.67 (30.943) | 6.40 (20.073) | 7.55 (26.095)
Hemoglobin at Week 52/Baseline [Mean (Standard Deviation); unit: g/dL] | 13.00 (1.405) | 12.81 (1.305) | 12.91 (1.356)
Index uterine fibroid volume at Week 52/Baseline [Mean (Standard Deviation); unit: cm^3] — Population: The data was reported for participants analyzed for each parameter
  cm^3
    number analyzed (Participants) | 115 | 112 | 227
    (all) | 40.06 (59.093) | 70.36 (142.863) | 55.01 (109.619)
Uterine Volume at Week 52/Baseline [Mean (Standard Deviation); unit: cm^3] | 274.95 (201.122) | 324.98 (309.228) | 299.75 (261.001)
UFS-QoL Bleeding and Pelvic Discomfort (BPD) Scale Score at Week 52/Baseline [Mean (Standard Deviation); unit: score on a scale] — The BPD Scale is derived from the UFS-QoL Symptoms Scale and was completed by participants on a paper at the study site before other study procedures. It consists of 3 symptoms proximal to uterine fibroids: Heavy bleeding during your menstrual period; Passing blood clots during your menstrual period; Feeling tightness or pressure in your pelvic area. To calculate the score, the 3 items are summed and transformed to a normalized score (range 0 to 100). Higher scores indicate greater severity and lower scores indicate minimal severity (high scores = bad).
  score on a scale | 10.51 (17.138) | 15.12 (24.027) | 12.79 (20.921)
UFS-QoL Symptom Severity Score at Week 52/Baseline [Mean (Standard Deviation); unit: score on a scale] — The UFS-QoL Symptom Severity scale assesses symptom severity in patients with uterine fibroids and was completed by participants on a paper at the study site before other study procedures. It consists of 8-items scored on a 5-point scale ranging from "not at all" to "a very great deal." To calculate the score, the 8 items are summed and transformed to a normalized score (range 0 to 100). Higher scores indicate greater severity and lower scores indicate minimal severity (high scores = bad).
  score on a scale | 14.62 (18.346) | 18.36 (22.659) | 16.47 (20.636)
Uterine Fibroid Symptom and Health-Related Quality of Life (UFS-QoL) Total Score at Week 52/Baseline [Mean (Standard Deviation); unit: scores on a scale] — The UFS-QoL assesses symptom severity and quality-of-life in patients with uterine fibroids and was completed by participants on a paper at the study site before other study procedures. Total score includes the 8-item symptom severity scale and 29-item QoL scale. All are scored on a 5-point Likert scale; symptom severity items range from "not at all" to "a very great deal" and QoL items range from "none of the time" to "all of the time." The values for each scale are summed and transformed to normalized scores (range 0 to 100). Higher scores indicate better health-related QoL (high = good).
  scores on a scale | 86.07 (18.566) | 81.06 (21.971) | 83.59 (20.435)
Patient Global Assessment (PGA) for uterine fibroid-related function at Week 52/Baseline [Count of Participants; unit: Participants]
  No limitation at all | 94 | 94 | 188
  Mild limitation | 12 | 10 | 22
  Moderate limitation | 4 | 5 | 9
  Quite a bit of limitation | 2 | 2 | 4
  Extreme limitation | 3 | 2 | 5
PGA for uterine fibroid-related symptom at Week 52/Baseline [Count of Participants; unit: Participants]
  Not severe | 99 | 97 | 196
  Mildly severe | 6 | 7 | 13
  Moderately severe | 6 | 4 | 10
  Very severe | 2 | 2 | 4
  Extremely severe | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage Of Participants Who Maintained MBL Volume Of <80 Milliliters (mL) At Week 76 During The Randomized Treatment Period
Description: MBL volume is measured using the alkaline hematin method. The method involves pummeling used feminine products in a 5% sodium hydroxide solution, which leads to the conversion of hemoglobin to alkaline hematin. The volume of MBL is measured in mL and a blood loss of 80 mL or more per cycle is considered diagnostic of heavy menstrual bleeding. The sustained responder rate was calculated as the Kaplan-Meier estimate of the cumulative probability of MBL volume < 80 mL through Week 76 using the Kaplan-Meier method.
Time Frame: Week 52/Baseline up to Week 76
Population: mITT population: all participants randomized to treatment who had taken at least 1 dose of study treatment (relugolix plus E2/NETA or placebo).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 115 | 113
percentage of participants | 78.43 [69.33 to 85.12] | 15.08 [8.91 to 22.76]
Statistical Analysis 1: Comparison: Relugolix Plus E2/NETA (Group A) vs Placebo (Group B); The primary efficacy analysis was the comparison of the relugolix plus E2/NETA group with the placebo group with respect to responder rate; Test type: Other — Chi-square test was used for the comparison between relugolix plus E2/NETA group and placebo group; p < 0.0001, Log-Log transformation — P-value was based on the stratified test statistics via log-log transformation of the difference in survival curve at a fixed time point stratified by pivotal study baseline MBL volume and duration of prior exposure to relugolix; Log-Log transformation of survival curve based on stratified Kaplan-Meier analysis; Treatment difference = 63.36, 95% CI 2-sided [52.85 to 73.86] — The 95% confidence interval (CI) of treatment difference was calculated via linear transformation of the difference in survival function with pooled variance

2. Secondary Outcome: Time To MBL Volume ≥80 mL During The Randomized Treatment Period
Description: MBL volume is measured using the alkaline hematin method. The method involves pummeling used feminine products in a 5% sodium hydroxide solution, which leads to the conversion of hemoglobin to alkaline hematin. The volume of MBL is measured in mL and a blood loss of 80 mL or more per cycle is considered diagnostic of heavy menstrual bleeding.
Time Frame: From Week 52/Baseline through Week 104
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 115 | 113
weeks | NA [NA to NA] — Median time to relapse was not reached due to the small number of participants with events (fewer than 50% of participants relapsed) | 5.9 [5.4 to 6.3]
Statistical Analysis 1: Comparison: Relugolix Plus E2/NETA (Group A) vs Placebo (Group B); Test type: Other — Stratified log-rank test was used for the comparison between relugolix plus E2/NETA group and placebo group; p < 0.0001, Log Rank — P-value for comparison of relugolix plus E2/NETA to placebo was based on the stratified log-rank test; Hazard Ratio (HR) = 0.13, 95% CI 2-sided [0.08 to 0.20] — Hazard ratio (95% CI) of relugolix plus E2/NETA to placebo was based on a proportional hazard model stratified by pivotal study baseline MBL volume (<225 mL or ≥225 mL) and duration of prior exposure to relugolix (28 weeks or 52 weeks)

3. Secondary Outcome: Percentage Of Participants Who Maintained MBL Volume Of <80 mL At Week 104 During The Randomized Treatment Period
Description: MBL volume is measured using the alkaline hematin method. The method involves pummeling used feminine products in a 5% sodium hydroxide solution, which leads to the conversion of hemoglobin to alkaline hematin. The volume of MBL is measured in mL and a blood loss of 80 mL or more per cycle is considered diagnostic of heavy menstrual bleeding. The sustained responder rate was calculated as the Kaplan-Meier estimate of the cumulative probability of MBL volume < 80 mL through Week 104 using the Kaplan-Meier method.
Time Frame: Week 52/Baseline up to Week 104
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 115 | 113
percentage of participants | 69.79 [59.72 to 77.80] | 11.75 [6.32 to 19.00]
Statistical Analysis 1: Comparison: Relugolix Plus E2/NETA (Group A) vs Placebo (Group B); Test type: Other — Chi-square test was used for the comparison between relugolix plus E2/NETA group and placebo group; p < 0.0001, Log-Log transformation — [p-value comment as in outcome 1, analysis 1]; Log-Log transformation of survival curve based on stratified Kaplan-Meier analysis; Treatment difference = 58.04, 95% CI 2-sided [46.97 to 69.11] — The 95% CI of treatment difference was calculated via linear transformation of the difference in survival function with pooled variance

4. Secondary Outcome: Percentage Of Participants Achieving Or Maintaining Amenorrhea At Week 76 During The Randomized Treatment Period
Description: Assessed using participant daily diary and MBL volume measured using the alkaline hematin method. Participants were deemed to be amenorrhoeic if one of the following criteria was met: No feminine products returned due to reported amenorrhea, or No feminine products returned due to reported spotting or feminine product collection with a negligible observed MBL volume (<5 mL) coupled with other data indicating infrequent non-cyclic bleeding/spotting. If no feminine product collection because participant failed to collect used products per protocol or due to "Other" reason, the amenorrhea status was set to missing. Missing responses for menstrual bleeding questions in the paper diary were treated as "No Bleeding" if paper diary entry/compliance rate was >70%.
Time Frame: Week 76
Population: mITT population: all participants randomized to treatment who had taken at least 1 dose of study treatment (relugolix plus E2/NETA and placebo).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 115 | 113
percentage of participants | 57.39 [47.83 to 66.56] | 13.27 [7.62 to 20.95]
Statistical Analysis 1: Comparison: Relugolix Plus E2/NETA (Group A) vs Placebo (Group B); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value for difference between relugolix plus E2/NETA and placebo is based on Cochran-Mantel-Haenszel test stratified by pivotal study baseline MBL volume (<225 mL or ≥225 mL) and duration of prior exposure to relugolix (28 weeks or 52 weeks); Treatment difference = 44.12, 95% CI 2-sided [33.13 to 55.11] — Treatment difference is relugolix plus E2/NETA minus placebo. 95% CI for difference is based on the normal approximation

5. Secondary Outcome: Change From Week 52/Baseline To Week 76 In MBL Volume During The Randomized Treatment Period
Description: MBL volume is measured using the alkaline hematin method. The method involves pummeling used feminine products in a 5% sodium hydroxide solution, which leads to the conversion of hemoglobin to alkaline hematin. Participants with amenorrhea are assigned with an MBL value of 0 mL and participants with spotting are assigned with an MBL value of 4.99 mL. The volume of MBL is measured in mL and a blood loss of 80 mL or more per cycle is considered diagnostic of heavy menstrual bleeding.
Time Frame: Week 52/Baseline to Week 76
Population: mITT population: all participants randomized to treatment who had taken at least 1 dose of study treatment (relugolix E2/NETA or placebo). Number analyzed represents proportion of overall group with values at that time point.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 81 | 17
mL | 6.6 (42.80) | 11.5 (27.45)

6. Secondary Outcome: Change From Week 52/Baseline To Week 104 In MBL Volume During The Randomized Treatment Period
Description: as for outcome 5
Time Frame: Week 52/Baseline to Week 104
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 63 | 8
mL | 2.1 (28.85) | 3.9 (10.92)

7. Secondary Outcome: Percentage Change From Week 52/Baseline To Week 76 In MBL Volume During The Randomized Treatment Period
Description: as for outcome 5
Time Frame: Week 52/Baseline to Week 76
Population: mITT population: all randomized participants who had taken at least 1 dose of study treatment. The % change from Week 52 in MBL volume was only available when Week 52 MBL volume is > 0 mL and post-Week 52 MBL volumes were available. The majority of mITT participants had MBL volume of 0 mL at Week 52/Baseline (92/115 in Group A and 89/113 in Group B). Number analyzed represents proportion of mITT population with MBL volume > 0 mL at Week 52 and values at each time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 14 | 2
percent change | 652.0 (1759.37) | 55.0 (219.15)

8. Secondary Outcome: Percentage Change From Week 52/Baseline To Week 104 In MBL Volume During The Randomized Treatment Period
Description: as for outcome 5
Time Frame: Week 52/Baseline to Week 104
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 8 | 0
percent change | -42.0 (48.80) |

9. Secondary Outcome: Percentage Of Participants Achieving Or Maintaining Amenorrhea At Week 104 During The Randomized Treatment Period
Description: Assessed using participant daily diary and MBL volume measured using the alkaline hematin method. Participants were deemed to be amenorrhoeic if one of the following criteria was met: No feminine products returned due to reported amenorrhea or no feminine products returned due to reported spotting or feminine product collection with a negligible observed MBL volume (<5 mL) coupled with other data indicating infrequent non-cyclic bleeding/spotting. If no feminine product collection because participant failed to collect used products per protocol or due to "Other" reason, the amenorrhea status was set to missing. Missing responses for menstrual bleeding questions in the paper diary were treated as "No Bleeding" if paper diary entry/compliance rate was >70%.
Time Frame: Week 104
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 115 | 113
percentage of patients | 58.26 [48.70 to 67.39] | 10.62 [5.61 to 17.82]

10. Secondary Outcome: Percentage Of Participants Who Responded (MBL Volume <80 mL) To Retreatment During The Retreatment Period
Description: as for outcome 2
Time Frame: From Initiation of Retreatment to Week 104
Population: Retreatment population: comprised participants in the mITT population from both treatment groups whose MBL volume reached ≥ 80 mL during the randomized treatment period and who started retreatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 26 | 89
percentage of participants | 96.15 [80.36 to 99.90] | 97.75 [92.12 to 99.73]

11. Secondary Outcome: Percentage Of Participants Whose Menses Had Resumed During The Randomized Treatment Period
Description: Participants who were previously amenorrhoeic were deemed to resume menses according to the following rules: MBL volume of collected feminine product was ≥5 mL; MBL volume of collected feminine product was <5 mL; however, there were more than 5 days and more than 3 consecutive days of bleeding with feminine product use during the visit; no feminine products were returned because the participant failed to collect used products per protocol; however, there were more than 5 days and more than 3 consecutive days of bleeding with feminine product use during the visit; or no feminine products were returned due to other reasons that indicated menstruation had occurred; also, there were more than 5 days and more than 3 consecutive days of bleeding with feminine product use during the visit.
Time Frame: Week 52/Baseline to Week 76 and Week 104
Population: mITT population who was amenorrhoeic at Week 52/Baseline: all participants randomized to treatment who had taken at least 1 dose of study treatment (relugolix plus E2/NETA or placebo) and who were amenorrhoeic at Week 52/Baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 92 | 89
percentage of participants
  Week 76 | 35.29 [26.14 to 46.48] | 91.54 [84.33 to 96.28]
  Week 104 | 41.12 [31.22 to 52.75] | 92.75 [85.86 to 97.04]

12. Secondary Outcome: Time To Resumption Of Menses For Participants Who Were Amenorrhoeic At Week 52/Baseline During The Randomized Treatment Period
Description: Assessed using participant daily diary. Participants were deemed to be amenorrhoeic if one of the following criteria was met: No feminine products returned due to reported amenorrhea, or No feminine products returned due to reported spotting or feminine product collection with a negligible observed MBL volume (<5 mL) coupled with other data indicating infrequent non-cyclic bleeding/spotting. If no feminine product collection because participant failed to collect used products per protocol or due to "Other" reason, the amenorrhea status was set to missing. Missing responses for menstrual bleeding questions in the paper diary were treated as "No Bleeding" if paper diary entry/compliance rate was >70%.
Time Frame: Week 52/Baseline up to Week 104
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 92 | 89
weeks | NA [42.6 to NA] — Median time to menses resumption was not reached as <50% of participants did not resume menses within the 52-week randomized treatment period. | 5.4 [5.0 to 5.9]

13. Secondary Outcome: Change From Week 52/Baseline In Hemoglobin Concentration During The Randomized Treatment Period
Description: Blood samples were collected from participants for hemoglobin measurements in accordance with the specified time points.
Time Frame: Week 52/Baseline to Week 76
Population: mITT population: all participants randomized to treatment who had taken at least 1 dose of study treatment (relugolix plus E2/NETA or placebo). Number analyzed represents proportion of overall group with values at that time point.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 81 | 20
g/dL | 0.3 (0.96) | -0.1 (1.10)

14. Secondary Outcome: Change From Week 52/Baseline In Hemoglobin Concentration During The Randomized Treatment Period
Description: Blood samples were collected from participants for hemoglobin measurements in accordance with the specified time points.
Time Frame: Week 52/Baseline to Week 104
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 59 | 8
g/dL | 0.3 (1.03) | -0.2 (1.36)

15. Secondary Outcome: Percentage Of Participants With MBL Volume Of ≥80 mL At Week 76 And Week 104 During the Randomized Treatment Period
Description: as for outcome 2
Time Frame: From Week 52/Baseline to Week 76 and Week 104
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 115 | 113
percentage of participants
  At Week 76 | 21.57 [14.88 to 30.67] | 84.92 [77.24 to 91.09]
  At Week 104 | 30.21 [22.20 to 40.28] | 88.25 [81.00 to 93.68]

16. Secondary Outcome: Percent Change From Week 52/Baseline In Hemoglobin Concentration During The Randomized Treatment Period
Description: Blood samples were collected from participants for hemoglobin measurements in accordance with the specified time points.
Time Frame: Week 52/Baseline to Week 64
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 97 | 72
percent change | 1.3 (6.75) | -4.3 (8.53)

17. Secondary Outcome: Percent Change From Week 52/Baseline In Hemoglobin Concentration During The Randomized Treatment Period
Description: Blood samples were collected from participants for hemoglobin measurements in accordance with the specified time points.
Time Frame: Week 52/Baseline to Week 76
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 81 | 20
percent change | 2.8 (8.30) | -0.8 (9.10)

18. Secondary Outcome: Percent Change From Week 52/Baseline In Hemoglobin Concentration During The Randomized Treatment Period
Description: Blood samples were collected from participants for hemoglobin measurements in accordance with the specified time points.
Time Frame: Week 52/Baseline to Week 104
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 59 | 8
percent change | 2.3 (8.94) | -0.7 (10.65)

19. Secondary Outcome: Percentage Of Participants Who Had Hemoglobin Level ≤10.5 g/dL Over Time During The Randomized Treatment Period
Description: Blood samples were collected from participants for hemoglobin measurements in accordance with the specified time points.
Time Frame: Week 52/Baseline to Week 76
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 81 | 20
percentage of participants | 4.94 [1.36 to 12.16] | 10.00 [1.23 to 31.70]

20. Secondary Outcome: Percentage Of Participants Who Had Hemoglobin Level ≤10.5 g/dL Over Time During The Randomized Treatment Period
Description: Blood samples were collected from participants for hemoglobin measurements in accordance with the specified time points.
Time Frame: Week 52/Baseline to Week 104
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 59 | 8
percentage of participants | 5.08 [1.06 to 14.15] | 0 [0 to 36.94]

21. Secondary Outcome: Percentage Of Participants Who Had Hemoglobin Level <11.6 g/dL Over Time During The Randomized Treatment Period
Description: Blood samples were collected from participants for hemoglobin measurements in accordance with the specified time points.
Time Frame: Week 52/Baseline to Week 76
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 81 | 20
percentage of participants | 6.17 [2.03 to 13.82] | 15.00 [3.21 to 37.89]

22. Secondary Outcome: Percentage Of Participants Who Had Hemoglobin Level <11.6 g/dL Over Time During The Randomized Treatment Period
Description: Blood samples were collected from participants for hemoglobin measurements in accordance with the specified time points.
Time Frame: Week 52/Baseline to Week 104
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 59 | 8
percentage of participants | 6.78 [1.88 to 16.46] | 25.00 [3.19 to 65.09]

23. Secondary Outcome: Change From Week 52/Baseline In Short Form 36v2 (SF-36v2) Domain During The Randomized Treatment Period
Description: The Short-Form Health Survey Standard (SF-36) is a validated, 36-item questionnaire, assessing general overall quality of life and was completed by participants on paper before other study procedures were performed, except for at the Week 52/Baseline visit, which was completed after eligibility for this study was confirmed and all Week 52 procedures for the long-term extension study were completed. Scores are calculated for each domain and 2 summary scores - a physical component summary score (Domains [number of items]: Physical Functioning [10], Role-Physical [4], Bodily Pain [2], General Health [5]), a mental component summary score (Domains [number of items]: Vitality [4], Social Functioning [2], Role-Emotional [3], and Mental Health [5]), and reported Health Transition [1]. Individual domain and component summary scores range from 0 to 100. Higher scores indicate higher health-related quality of life.
Time Frame: Week 52/Baseline to Week 76
Population: mITT population: all participants randomized to treatment who had taken at least 1 dose of study treatment (relugolix plus E2/NETA or placebo). Number analyzed represents proportion of overall group with values for that measure at that time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 85 | 21
score on a scale
  Physical Functioning | 1.1 (4.24) | -2.3 (5.16)
  Role-Physical | 0.3 (4.80) | -1.2 (4.75)
  Bodily Pain | 0.6 (8.02) | -0.3 (9.78)
  General Health | 0 (6.68) | -3.1 (6.81)
  Vitality | 0.5 (7.87) | 0.4 (8.83)
  Social Functioning | -0.2 (7.85) | -2.9 (6.65)
  Role-Emotional | 0.6 (7.38) | -1.0 (7.23)
  Mental Health | 0.5 (8.30) | -1.0 (9.98)

24. Secondary Outcome: Change From Week 52/Baseline In Short Form 36v2 (SF-36v2) Domain During The Randomized Treatment Period
Description: as for outcome 23
Time Frame: Week 52/Baseline to Week 104
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 64 | 8
score on a scale
  Physical Functioning | 0.5 (5.44) | 0.5 (2.23)
  Role-Physical: number analyzed (Participants) | 63 | 8
  Role-Physical | -0.5 (6.49) | -0.6 (2.88)
  Bodily Pain | 1.9 (7.36) | 1.7 (8.42)
  General Health | -0.6 (5.67) | -5.5 (7.72)
  Vitality | 0.5 (7.53) | 3.0 (8.84)
  Social Functioning | -0.4 (7.85) | -0.6 (3.21)
  Role-Emotional: number analyzed (Participants) | 63 | 8
  Role-Emotional | -0.2 (7.32) | -3.9 (6.29)
  Mental Health | -0.8 (7.34) | 2.9 (9.83)

25. Secondary Outcome: Change From Week 52/Baseline In SF-36v2 Summary Component Scores During The Randomized Treatment Period
Description: The Short-Form Health Survey Standard (SF-36) is a validated, 36-item questionnaire, assessing general overall quality of life and was completed by participants on paper before other study procedures were performed, except for at the Week 52/Baseline visit, which was completed after eligibility for this study was confirmed and all Week 52 procedures for the long-term extension study were completed. Scores are calculated for each domain and 2 summary scores - a physical component summary (PCS) score (Domains [number of items]: Physical Functioning [10], Role-Physical [4], Bodily Pain [2], General Health [5]), a mental component summary (MCS) score (Domains [number of items]: Vitality [4], Social Functioning [2], Role-Emotional [3], and Mental Health [5]), and reported Health Transition [1]. Individual domain and component summary scores range from 0 to 100. Higher scores indicate higher health-related quality of life.
Time Frame: Week 52/Baseline to Week 76
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 85 | 21
score on a scale
  PCS | 0.6 (4.89) | -1.8 (6.00)
  MCS | 0.2 (7.93) | -0.8 (7.70)

26. Secondary Outcome: Change From Week 52/Baseline In SF-36v2 Summary Component Scores During The Randomized Treatment Period
Description: as for outcome 25
Time Frame: Week 52/Baseline to Week 104
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 63 | 8
score on a scale
  PCS | 0.8 (5.18) | -0.6 (4.04)
  MCS | -0.8 (6.65) | 0.1 (7.71)

27. Secondary Outcome: Categorical Change From Week 52/Baseline In PGA For Uterine Fibroid-related Function During The Randomized Treatment Period
Description: The PGA for function is a 1-item questionnaire designed to assess participant's impression of the impact on their function related to uterine fibroids affected their usual activities and was completed on paper. The PGA for function was evaluated using a 5-point Likert scale (1 = No limitation at all; 5 = Extreme limitation) with higher numbers representing worse results. Endpoint values represent the worsening of function (deterioration), improvement of function (improvement), or no change by category at each time point. For example, a 4-category deterioration represents a change from 1 (No limitation at all) to 5 (Extreme limitation) and a 4-category improvement represents a change from 5 (Extreme limitation) to 1 (No limitation at all).
Time Frame: Week 52/Baseline to Week 76
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 86 | 21
Participants
  4 Category deterioration | 0 | 0
  3 Category deterioration | 2 | 0
  2 Category deterioration | 4 | 3
  1 Category deterioration | 8 | 3
  No change | 63 | 14
  1 Category improvement | 5 | 1
  2 Category improvement | 2 | 0
  3 Category improvement | 1 | 0
  4 Category improvement | 1 | 0

28. Secondary Outcome: Categorical Change From Week 52/Baseline In PGA For Uterine Fibroid-related Function During The Randomized Treatment Period
Description: as for outcome 27
Time Frame: Week 52/Baseline to Week 104
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 65 | 8
Participants
  4 Category deterioration | 0 | 0
  3 Category deterioration | 0 | 0
  2 Category deterioration | 3 | 0
  1 Category deterioration | 4 | 1
  No change | 54 | 7
  1 Category improvement | 2 | 0
  2 Category improvement | 1 | 0
  3 Category improvement | 0 | 0
  4 Category improvement | 1 | 0

29. Secondary Outcome: Categorical Change From Week 52/Baseline In PGA For Uterine Fibroid-related Symptoms During The Randomized Treatment Period
Description: The PGA for symptoms is a 1-item questionnaire designed to assess participant's impression of the severity of their symptoms related to uterine fibroids and was completed on paper. The PGA for symptoms was evaluated using a 5-point Likert scale (1 = Not severe; 5 = Extremely severe) with higher numbers representing worse results. Endpoint values represent the worsening of symptoms (deterioration), improvement of symptoms (improvement), or no change by category at each time point. For example, a 4-category deterioration represents a change from 1 (Not severe) to 5 (Extremely severe) and a 4-category improvement represents a change from 5 (Extremely severe) to 1 (Not severe).
Time Frame: Week 52/Baseline to Week 76
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 86 | 21
Participants
  4 Category deterioration | 0 | 0
  3 Category deterioration | 1 | 1
  2 Category deterioration | 4 | 3
  1 Category deterioration | 8 | 3
  No change | 63 | 13
  1 Category improvement | 5 | 0
  2 Category improvement | 4 | 1
  3 Category improvement | 0 | 0
  4 Category improvement | 1 | 0

30. Secondary Outcome: Categorical Change From Week 52/Baseline In PGA For Uterine Fibroid-related Symptoms During The Randomized Treatment Period
Description: as for outcome 29
Time Frame: Week 52/Baseline to Week 104
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 65 | 8
Participants
  4 Category deterioration | 0 | 0
  3 Category deterioration | 1 | 0
  2 Category deterioration | 1 | 0
  1 Category deterioration | 0 | 1
  No change | 58 | 7
  1 Category improvement | 2 | 0
  2 Category improvement | 2 | 0
  3 Category improvement | 0 | 0
  4 Category improvement | 1 | 0

31. Secondary Outcome: Change From Week 52/Baseline In The Work Productivity Activity Impairment - Percent Work Time Missed Due to Uterine Fibroids (WPAI-UF) Scores During The Randomized Treatment Period
Description: The WPAI-UF is a validated instrument used to measure self-reported absenteeism, presenteeism, and daily activity impairment attributed to uterine fibroids. The WPAI-UF was to be completed on a paper questionnaire and participants were to answer these questions.
  Percent work time missed due to uterine fibroids was calculated from hours missed due to uterine fibroids divided by the sum of hours missed due to uterine fibroids plus hours actually worked. This value was then multiplied by 100 to get a percentage. The WPAI-UF outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity due to uterine fibroids, that is, worse outcomes.
Time Frame: Week 52/Baseline up to Week 76
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage score
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 62 | 13
percentage score | 0.7 (10.22) | 3.9 (13.85)

32. Secondary Outcome: Change From Week 52/Baseline In The Work Productivity Activity Impairment - Percent Work Time Missed Due to Uterine Fibroids (WPAI-UF) Scores During The Randomized Treatment Period
Description: as for outcome 31
Time Frame: Week 52/Baseline up to Week 104
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage score
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 48 | 5
percentage score | 0.5 (8.50) | 0 (0)

33. Secondary Outcome: Change From Week 52/Baseline In The Work Productivity Activity Impairment - Percent Impairment While Working Due to Uterine Fibroids (WPAI-UF) Scores During The Randomized Treatment Period
Description: The WPAI-UF is a validated instrument used to measure self-reported absenteeism, presenteeism, and daily activity impairment attributed to uterine fibroids. The WPAI-UF was to be completed on a paper questionnaire and participants were to answer these questions.
  Percent impairment while working due to uterine fibroid symptoms was calculated by taking the reported value from 1 (no effect) to 10 (completely prevented work) and dividing by 10. This value was then multiplied by 100 to get a percentage. The WPAI-UF outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity due to uterine fibroids, that is, worse outcomes.
Time Frame: Week 52/Baseline up to Week 76
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage score
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 70 | 17
percentage score | -1.1 (16.20) | 1.8 (15.90)

34. Secondary Outcome: Change From Week 52/Baseline In The Work Productivity Activity Impairment - Percent Impairment While Working Due to Uterine Fibroids (WPAI-UF) Scores During The Randomized Treatment Period
Description: as for outcome 33
Time Frame: Week 52/Baseline up to Week 104
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage score
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 54 | 6
percentage score | 0 (15.17) | 5.0 (12.25)

35. Secondary Outcome: Change From Week 52/Baseline In The Work Productivity Activity Impairment - Percent Overall Work Impairment Due to Uterine Fibroids (WPAI-UF) Scores During The Randomized Treatment Period
Description: The WPAI-UF is a validated instrument used to measure self-reported absenteeism, presenteeism, and daily activity impairment attributed to uterine fibroids. The WPAI-UF was to be completed on a paper questionnaire and participants were to answer these questions.
  Percent overall work impairment due to uterine fibroid symptoms was calculated from the work time missed due to uterine fibroids plus the value calculated from 1 minus the work time missed value multiplied by the value for impairment while working due to uterine fibroids. This value was then multiplied by 100 to get a percentage. The WPAI-UF outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity due to uterine fibroids, that is, worse outcomes.
Time Frame: Week 52/Baseline up to Week 76
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage score
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 62 | 13
percentage score | -0.8 (20.05) | 3.2 (10.56)

36. Secondary Outcome: Change From Week 52/Baseline In The Work Productivity Activity Impairment - Percent Overall Work Impairment Due to Uterine Fibroids (WPAI-UF) Scores During The Randomized Treatment Period
Description: as for outcome 35
Time Frame: Week 52/Baseline up to Week 104
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage score
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 48 | 5
percentage score | 0.6 (19.13) | 6.0 (13.42)

37. Secondary Outcome: Change From Week 52/Baseline In The Work Productivity Activity Impairment - Percent Activity Impairment Due to Uterine Fibroids (WPAI-UF) Scores During The Randomized Treatment Period
Description: The WPAI-UF is a validated instrument used to measure self-reported absenteeism, presenteeism, and daily activity impairment attributed to uterine fibroids. The WPAI-UF was to be completed on a paper questionnaire and participants were to answer these questions.
  Percent activity impairment due to uterine fibroid symptoms was calculated by taking the reported value from 1 (no effect) to 10 (completely prevented activity) and dividing by 10. This value was then multiplied by 100 to get a percentage. The WPAI-UF outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity due to uterine fibroids, that is, worse outcomes.
Time Frame: Week 52/Baseline up to Week 76
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage score
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 85 | 20
percentage score | -0.5 (21.10) | 4.5 (19.32)

38. Secondary Outcome: Change From Week 52/Baseline In The Work Productivity Activity Impairment - Percent Activity Impairment Due to Uterine Fibroids (WPAI-UF) Scores During The Randomized Treatment Period
Description: The WPAI-UF is a validated instrument used to measure self-reported absenteeism, presenteeism, and daily activity impairment attributed to uterine fibroids. The WPAI-UF was to be completed on a paper questionnaire and participants were to answer these questions.
  Percent activity impairment due to uterine fibroid symptoms was calculated by taking the reported value from 1 (no effect) to 10 (completely prevented work) and dividing by 10. This value was then multiplied by 100 to get a percentage. The WPAI-UF outcomes are expressed as impairment percentages (0 to 100%), with higher numbers indicating greater impairment and less productivity due to uterine fibroids, that is, worse outcomes.
Time Frame: Week 52/Baseline up to Week 104
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage score
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 64 | 8
percentage score | -1.3 (18.90) | 5.0 (10.69)

39. Secondary Outcome: Change From Week 52/Baseline In The UFS-QoL Bleeding And Pelvic Discomfort Score During The Randomized Treatment Period
Description: Assessed using the UFS-QOL which is a validated instrument used to evaluate symptom severity and quality of life in participants with uterine fibroids. The UFS-QoL was completed on a paper questionnaire and participants were to answer the following questions: heavy bleeding during your menstrual period (Question 1), passing blood clots during your menstrual period (Question 2), and feeling tightness or pressure in your pelvic area (Question 5). Items are scored on a 5-point scale, ranging from "not at all" to "a very great deal." A summed score was created for questions 1, 2, and 5 and transformed to a normalized score with a range of possible values from 0 to 100, where a higher score was indicative of greater distress and a lower score of less distress (high scores = bad).
Time Frame: Week 52/Baseline to Week 76
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 86 | 21
score on a scale | 3.4 (20.27) | 17.5 (24.99)

40. Secondary Outcome: Change From Week 52/Baseline In The UFS-QoL Bleeding And Pelvic Discomfort Score During The Randomized Treatment Period
Description: as for outcome 39
Time Frame: Week 52/Baseline to Week 104
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 65 | 8
score on a scale | -0.5 (17.85) | -6.3 (43.36)

41. Secondary Outcome: Original: Change From Week 52/Baseline In The UFS-QoL Symptom Severity Score During The Randomized Treatment Period
Description: Assessed using the UFS-QOL, which is a validated instrument used to evaluate symptom severity and quality of life in participants with uterine fibroids. The UFS-QoL was completed on a paper questionnaire and participants were to answer these questions. Items are scored on a 5-point scale, ranging from "not at all" to "a very great deal." A summed score was created for questions 1 through 8 and transformed to a normalized score with a range of possible values from 0 to 100, where a higher score was indicative of greater symptom severity and a lower score of lower symptom severity (negative score = improvement).
Time Frame: Week 52/Baseline to Week 76
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 86 | 21
score on a scale | 2.2 (18.16) | 14.1 (21.07)

42. Secondary Outcome: New: Change From Week 52/Baseline In The UFS-QoL Symptom Severity Score During The Randomized Treatment Period
Description: as for outcome 41
Time Frame: Week 52/Baseline to Week 104
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 65 | 8
score on a scale | 0.1 (15.94) | -4.3 (42.22)

43. Secondary Outcome: Change From Week 52/Baseline In The UFS-QoL Score by Health-Related Quality Of Life Subscale And Total Scores During The Randomized Treatment Period
Description: Assessed using the UFS-QOL which, is a validated instrument used to evaluate symptom severity and quality of life in participants with uterine fibroids. Items are scored on a 5-point scale, ranging from "none of the time" to "all of the time." The UFS-QoL was completed on a paper questionnaire and participants were to answer these questions. Questions 9 through 37 were used to calculate the total scores and the following subscales: concern, activities, revised activities, energy/mood, control, self-conscious, and sexual function. All raw scores are transformed to normalized scores with a range of possible values from 0 to 100. A positive score indicates improvement.
Time Frame: Week 52/Baseline to Week 76
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 86 | 21
score on a scale
  Concern | -2.4 (24.38) | -13.6 (27.76)
  Activities | -1.7 (17.46) | -11.7 (26.10)
  Revised activities | -2.3 (18.66) | -13.3 (27.13)
  Energy/mood | -0.1 (17.30) | -3.9 (23.69)
  Control | 0.2 (15.60) | -3.6 (23.03)
  Self-conscious | 0 (21.66) | -11.5 (16.77)
  Sexual function | 1.0 (28.77) | -16.7 (43.72)
  Total Score | -0.8 (16.79) | -9.1 (22.37)

44. Secondary Outcome: Change From Week 52/Baseline In The UFS-QoL Score by Health-Related Quality Of Life Subscale And Total Scores During The Randomized Treatment Period
Description: as for outcome 43
Time Frame: Week 52/Baseline to Week 104
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 65 | 8
score on a scale
  Concern | 2.2 (21.45) | 11.9 (41.40)
  Activities | 0.9 (16.74) | 8.5 (42.00)
  Revised activities | 0.6 (16.02) | 7.5 (42.59)
  Energy/mood | 1.6 (17.41) | 8.0 (44.35)
  Control | 1.7 (15.19) | 9.4 (39.05)
  Self-conscious | -2.8 (19.94) | 3.1 (44.53)
  Sexual function | 0.8 (26.51) | 3.1 (52.08)
  Total Score | 1.1 (15.25) | 8.2 (42.12)

45. Secondary Outcome: Predose Concentration Of Estradiol At Week 56
Description: Blood samples were collected from participants for estradiol measurements and were analyzed using a standard clinical methodology. The change from Week 52/Baseline in estradiol concentration at Week 56 was presented in this outcome.
Time Frame: Week 52/Baseline and Week 56
Population: Safety population: all randomized participants who received at least 1 dose of study treatment. Overall number of participants analyzed represents proportion of overall group with values at that time point.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 88 | 75
pg/mL | 2.03 (31.605) | 62.54 (77.661)

46. Secondary Outcome: Participants With Adverse Events (AEs) As A Measure Of Safety And Tolerability
Description: Assessed by percentage of participants with AEs and serious AEs (SAEs). An AE was defined as any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product, whether or not related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; or a congenital anomaly/birth defect. Events of heavy menstrual bleeding were only reported if the event met criteria as an SAE. A summary of serious and all other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Week 52/Baseline up to Week 104
Population: Safety population: all randomized participants who received at least 1 dose of study treatment. Note: One patient who was randomized to the placebo group was inadvertently dispensed open-label study drug of which the patient took 1 dose of relugolix + E2/NETA. Thus, the patient was considered as part of the relugolix + E2/NETA group in the Safety Population only. This changes the Group A population from 115 (mITT population) to 116 and the Group B population from 113 (mITT population) to 112.
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 116 | 112
Participants
  Any AEs | 68 | 72
  Leading to study treatment discontinuation | 2 | 3
  Leading to study treatment interruption | 1 | 0
  Related to study drug | 26 | 27
  Grade 3 or higher | 3 | 5
  Grade 3 or higher related to study drug | 0 | 2
  SAEs | 2 | 2
  Serious and related to study drug | 0 | 1
  Serious and leading to treatment discontinuation | 1 | 1
  Fatal outcome | 0 | 0

47. Secondary Outcome: Percent Change From Week 52/Baseline In BMD At Lumbar Spine (L1-L4)
Description: Assessed by dual-energy X-ray absorptiometry scan at the lumbar spine (L1-L4), total hip [presented separately], and femoral neck (same leg within each participant) [presented separately] at each designated timepoints. The least squares means and their 95% CI were based on analysis of covariance model with treatment, stratification factors, race as fixed factors, and age at Week 52/Baseline, Week 52/Baseline BMD value, and body mass index at Week 52/Baseline as covariates.
Time Frame: Week 52/Baseline to Week 104
Population: Safety population: all randomized participants who received at least 1 dose of study treatment. Note: 1 patient was randomized to placebo and inadvertently dispensed open-label study drug; the patient took 1 dose and was considered part of Group A in the Safety population only and is represented in the Overall Number of Participants Analyzed. Number analyzed by location/group represents proportion of the Safety population with values for that measure at that time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 79 | 79
percent change | 0.81 [0.20 to 1.41] | 0.10 [-0.52 to 0.71]

48. Secondary Outcome: Percent Change From Week 52/Baseline In BMD At Femoral Neck And Total Hip
Description: Assessed by dual-energy X-ray absorptiometry scan at the lumbar spine (L1-L4) [presented separately], total hip, and femoral neck (same leg within each participant) at each designated timepoints. The least squares means and their 95% CI were based on analysis of covariance model with treatment, stratification factors, race as fixed factors, and age at Week 52/Baseline, Week 52/Baseline BMD value, and body mass index at Week 52/Baseline as covariates.
Time Frame: Week 52/Baseline to Week 104
Population: as for outcome 47
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
Number analyzed (Participants) | 79 | 77
percent change
  Total Hip | 0.34 [-0.25 to 0.93] | -0.13 [-0.73 to 0.47]
  Femoral Neck | -0.19 [-1.14 to 0.77] | -0.76 [-1.74 to 0.21]

ADVERSE EVENTS:
Time Frame: Week 52/Baseline up to Week 104
Description: Safety population: all randomized participants who received at least 1 dose of study treatment.
  Note: One patient who was randomized to the placebo group was inadvertently dispensed open-label study drug of which the patient took 1 dose of relugolix + E2/NETA. Thus, the patient was considered as part of the relugolix + E2/NETA group in the Safety Population only. This changes the Group A population from 115 (mITT population) to 116 and the Group B population from 113 (mITT population) to 112.
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group B)
All-Cause Mortality (participants affected / at risk) | 0/116 | 0/112
Serious Adverse Events (participants affected / at risk) | 2/116 | 2/112
Other Adverse Events (participants affected / at risk) | 29/116 | 45/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Relugolix Plus E2/NETA (Group A) (N=116) | Placebo (Group B) (N=112)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myxoid liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transient global amnesia (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Relugolix Plus E2/NETA (Group A) (N=116) | Placebo (Group B) (N=112)
Nasopharyngitis (Infections and infestations) | 13 | 12
Headache (Nervous system disorders) | 8 | 5
Dysmenorrhoea (Reproductive system and breast disorders) | 2 | 8
Hot flush (Vascular disorders) | 2 | 8
Hypertension (Vascular disorders) | 2 | 6
Upper respiratory tract infection (Infections and infestations) | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-08-13): https://cdn.clinicaltrials.gov/large-docs/24/NCT03751124/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-15): https://cdn.clinicaltrials.gov/large-docs/24/NCT03751124/SAP_001.pdf